CLINICAL TRIAL: NCT05131542
Title: Development of a Measuring Instrument for the Evaluation of Hypotonia in Children With Down Syndrome
Brief Title: Assessment of Hypotonia in Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, María Guadalupe de Santos Moreno, Principal Investigator, Universidad de Murcia
Other Study IDs: 1999/2018
Record Dates: First submitted 2021-10-21; First posted 2021-11-23 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Muscle Hypotonia; Down Syndrome; Muscle, Floppy; CHILD Syndrome; Infant Floppy
MeSH Terms: conditions — Muscle Hypotonia; Down Syndrome; Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Down Syndrome: Children with down syndrome

SUMMARY:
Hypotonia is a common trait in infants with Down syndrome, resulting in pathologies and delays in gaining basic motor skills. There are no screenings available to aid in early diagnosis, therefore, the purpose of this study is to develop a way to test for hypotonia in children with Down syndrome.

DETAILED DESCRIPTION:
Hypotonia is usually diagnosed by observation and clinical assessment. Aiming to develop an instrument for early diagnosis, a systematic review was carried out which compiled characteristics and testing that are attributed to or used in the diagnosis of hypotonia. They were presented as an item group and a first stage was created and administered to 50 children with Down's Syndrome between the ages of 7 months to 8 years old. The study of the results showed which characteristics were really related to the convention and which were more affected by changing factors. Then a final scale was developed that met the expected requirements of validity and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer parents who have Infants with Down Syndrome Between the ages of 7 months to 8 years old

Exclusion Criteria:

* Other hypotonic syndromes

Ages: 7 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Down Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Quality assessment of items by homogeneity analysis. Statistical analysis was performed using the SPSS-21 program. | 1 month
  A study of homogeneity of the items was carried out to know if each item was measuring the same as the globality of the test. It was carried out by means of a reliability study of the statistics of each item compared to the total scale.
Analysis of the reliability of the scale | 1 month
  Reliability was measured by Cronbach's alpha. An interclass and inter-judge correlation analysis was performed
Content validity | 1 month
  It was done through expert judgment. It was reviewed by three physiotherapists with extensive experience in treating hypotonic children and those items directed to the orofacial complex were also agreed with an expert speech therapist.
Empirical validity. | 1 month
  The correlation between the graduation of hypotonia derived from the scale and the observational diagnosis estimated by the evaluator was analyzed. An ANOVA test was used to compare both diagnostic assessments.extensive experience in treating hypotonic children and those items directed to the orofacial complex were also agreed with an expert speech therapist.
Structural validity | In the process of analysis. 1 month to get results.
  Through an exploratory factor analysis. Factorial analysis was carried out using the FACTOR program.

SECONDARY OUTCOMES:
Descriptive analysis of the scale | 1 month
  Analyzing the values of standard deviation, mean, bias and kurtosis.
Frequency analysis of the items. | 1 month
  Frequency with which 0 (less hypotonia), 1 or 2 (greater hypotonia) each item of the scale has been scored.
Analysis of the scale items. | 1 month
  An analysis of standard deviation, mean, correlation and Cronbach's alpha was performed for each item that made up the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mª Guadalupe de Santos Moreno, MSc PT, Principal Investigator — Unicersity of Murcia; Antonia Gómez Conesa, PhD PT, Study Director — Unicersity of Murcia; José Antonio López Pina, PhD, Study Director — Unicersity of Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin K, Inman J, Kirschner A, Deming K, Gumbel R, Voelker L. Characteristics of hypotonia in children: a consensus opinion of pediatric occupational and physical therapists. Pediatr Phys Ther. 2005 Winter;17(4):275-82. doi: 10.1097/01.pep.0000186506.48500.7c. PMID 16357683
- [Background] Govender P, Joubert RWE. 'Toning' up hypotonia assessment: A proposal and critique. Afr J Disabil. 2016 May 26;5(1):231. doi: 10.4102/ajod.v5i1.231. eCollection 2016. PMID 28730054
- [Background] Goo M, Tucker K, Johnston LM. Muscle tone assessments for children aged 0 to 12 years: a systematic review. Dev Med Child Neurol. 2018 Jul;60(7):660-671. doi: 10.1111/dmcn.13668. Epub 2018 Feb 6. PMID 29405265
- [Background] Martin K, Kaltenmark T, Lewallen A, Smith C, Yoshida A. Clinical characteristics of hypotonia: a survey of pediatric physical and occupational therapists. Pediatr Phys Ther. 2007 Fall;19(3):217-26. doi: 10.1097/PEP.0b013e3180f62bb0. PMID 17700351
- [Background] Govender P, Joubert RWE. Evidence-Based Clinical Algorithm for Hypotonia Assessment: To Pardon the Errs. Occup Ther Int. 2018 Apr 24;2018:8967572. doi: 10.1155/2018/8967572. eCollection 2018. PMID 29853815
- [Background] Naidoo P, Joubert RW. Consensus on hypotonia via Delphi process. Indian J Pediatr. 2013 Aug;80(8):641-50. doi: 10.1007/s12098-013-1018-7. Epub 2013 May 17. PMID 23681830
- [Background] Reus L, van Vlimmeren LA, Staal JB, Janssen AJ, Otten BJ, Pelzer BJ, Nijhuis-van der Sanden MW. Objective evaluation of muscle strength in infants with hypotonia and muscle weakness. Res Dev Disabil. 2013 Apr;34(4):1160-9. doi: 10.1016/j.ridd.2012.12.015. Epub 2013 Feb 1. PMID 23380578
- [Background] Naidoo P. Development of an evidence-based clinical algorithm for practice in hypotonia assessment: a proposal. JMIR Res Protoc. 2014 Dec 5;3(4):e71. doi: 10.2196/resprot.3581. PMID 25485571
- See also: The American Academy for Cerebral Palsy and Developmental Medicine, develops a care pathway for therapeutic interventions for central hypotonia — http://www.aacpdm.org/publications/care-pathways/central-hypotonia